CLINICAL TRIAL: NCT03641092
Title: Evaluation of the Impact of the CenteringParenting Clinical Intervention on Kindergarten Readiness in Early Childhood
Brief Title: CenteringParenting Clinical Intervention on Kindergarten Readiness in Early Childhood
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Boston Medical Center (Other)
Collaborators: Centering Healthcare Institute (Other); Overdeck Family foundation (Other); Valhalla Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: H-37893
Record Dates: First submitted 2018-07-04; First posted 2018-08-21 (Actual); Last update posted 2025-12-01 (Actual); Status verified 2025-11

CONDITIONS: Parent-Child Relations; Parenting; Child Development; Child Behavior
Keywords: School readiness; Child development; Child behavior; Parenting behavior; CenteringParenting
MeSH Terms: conditions — Child Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Clinical Site (Experimental): 5 experimental clinical sites will receive the implementation of CenteringParenting assistance early. This arm will include the CenteringParenting intervention.
  Interventions: Behavioral: CenteringParenting Intervention
- Comparison Clinical Site (Active Comparator): 5 comparison clinical sites will receive Routine Well Child Care and CenteringParenting implementation assistance later and serve as control sites. This arm will include the Routine Well Child Care intervention.
  Interventions: Behavioral: Routine Well Child Care

INTERVENTIONS:
Behavioral: CenteringParenting Intervention — The CenteringParenting(CP) intervention includes group well child care visits during the first 24 months of life. Participants receive a journal with child safety, health and development information. The groups are co-led by a practitioner and support staff member. This bundled intervention supports healthy parent-child interactions and early learning through education and experiential learning within the well-child visit.
  Arms: Experimental Clinical Site
Behavioral: Routine Well Child Care — The Comparison Clinical Sites will receive the Routine Well Child Care standard individual clinical care. This clinic will receive delayed training in the CenteringParenting(CP) intervention approximately 3 months after the completion of recruitment at their study site [when recruited families will be ineligible for CenteringParenting groups that will start in control sites]. They will receive anticipatory guidance and handouts that are standard for the clinic.
  Arms: Comparison Clinical Site

SUMMARY:
Disparities in health begin in early childhood. Early life experiences influence brain development and have significant implications on future health and developmental outcomes. Low-income children are at greater risk of developmental delays in large part due to a lack of an enriched environment. Disparities in early childhood development increase risk for stunted academic achievement throughout the life course. Primary care is a universal exposure in early childhood and therefore is also a significant entry point for promoting optimal child development.

There is a need to provide effective, low-cost, and scalable interventions in primary care to support early childhood development.The CenteringParenting intervention is designed to reduce negative health and developmental outcomes within a model of group routine child health care. To date, there is no evidence of the benefits of the CenteringParenting intervention on school readiness, or improvements in parental behaviors that support optimal developmental milestones and achievement. The intent of this study is to determine the effectiveness of the CenteringParenting intervention on school readiness in early childhood, as measured by language development at 24 months, (in addition to health care utilization, child routine care maintenance, parenting stress, caregiver behaviors and attitudes).

DETAILED DESCRIPTION:
Children raised in environments with limited stimulation and lack of exposure to positive interactions are likely to have developmental delays in expressive and receptive language, vocabulary, social skills, behavior-all factors critical for school readiness. Children who enter kindergarten underprepared are more likely to struggle academically and experience lower school achievement, and ultimately impaired opportunities for economic and social mobility as adults.

The CenteringParenting intervention is designed to reduce negative health and developmental outcomes within a model of group routine child health care. This bundled intervention supports healthy parent-child interactions and early learning through education and experiential learning within a group well-child visit model. The intervention reduces social isolation and creates a community of support for caregivers, as well as utilizes a positive parenting approach to empowering parents with knowledge and skills to support optimal child development. The CenteringParenting intervention includes written materials provided at an annual clinical visit, as well as specific training for the facilitators/providers. To date, there is no research evidence of the benefits of the CenteringParenting intervention on school readiness, or improvements in parental behaviors that support optimal developmental milestones and achievement.

Study Design: A multi-site, cluster randomized controlled trial evaluating the impact of the CenteringParenting clinical intervention on kindergarten readiness, as measured by expressive and receptive language and vocabulary at 24 months of age.

Objective Hypothesis: Compared to those receiving standard routine health care, the CenteringParenting intervention will result in improved language development at age 2 years and increased parental behaviors to encourage reading, talking and playing.

Specific Aim 1: In a cluster randomized controlled trial, assess the effectiveness and implementation of the CenteringParenting intervention. Specific Aim 2: Evaluate the fidelity of the implementation of the CenteringParenting intervention. Specific Aim 3: Evaluate caregivers' experience and engagement with the CenteringParenting intervention model and explore the relation between degree of engagement and development stimulating behaviors.

Primary outcomes are: expressive and receptive language and vocabulary based on the MacArthur-Bates Communicative Development Inventory (CDI) and Preschool Language Scale-5 (PLS-5) 5th Edition Parent Questionnaire. The secondary outcome is: parental behavior based on the Stim-Q (a reliable and valid measure of cognitive stimulation provided in the home).

ELIGIBILITY:
Inclusion Criteria:

For participating practice sites

* Practice provides care to patients who are covered by public insurance and/or uninsured (no minimum threshold: all insurance types eligible)
* Practices have at least 3,000 primary care visits per year

For parent-child dyad

* Index child age must be 0-3 months
* Parent must be female
* Parent must be 18 years of age and older
* Parent and child must attend one of the 10 study clinical sites
* Parental consent
* Parent must be fluent in English or Spanish

Exclusion Criteria:

For participating practice sites

* Does not accept public insurance

For parent-child dyad

* Child born prior to 34 weeks gestation
* Child with chronic conditions known to affect neurodevelopment
* Child with a positive screen on the Children with Special Healthcare Needs screener

Max Age: 3 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 1200 (Estimated)
Dates: Start 2019-02-19 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Early language assessment at 12 months | 12 months
  Assess early language (vocabulary, comprehension, production, gestures and grammar) based on the MacArthur Communicative Development Inventories (CDI). The Words and Gestures short form (Level I) is comprised of a 89-word vocabulary checklist with separate columns for comprehension and production, appropriate for children 8-18 months. The score is assessed in the amount of correct answers and measured in percentiles, from <1th to 100th, depending on the child's age. Administered by research assistant to female guardian.
Early language assessment at 24 months | 24 months
  Assess early language (vocabulary, comprehension, production, gestures and grammar) based on the MacArthur Communicative Development Inventories (CDI). Two equivalent Words & Sentences versions (Level IIA and Level IIB) contain a 100-word productive vocabulary checklist and a question about combining words, appropriate for children 16-30 months. The score is assessed in the amount of correct answers and measured in percentiles, from <1th to 100th, depending on the child's age. Administered by research assistant to female guardian.
Receptive vocabulary assessment at 3 months | 3 months
  Assess Receptive vocabulary based on the Preschool Language Scale-5 (PLS-5) 5th Edition Parent Questionnaire. The scale accesses: Total language, auditory comprehension, expressive communication standard scores, growth scores, percentile ranks, language age equivalents. PLS-5 scores range anywhere from 40-160 with the mean being 100 and an SD of 15. Higher percentile ranks are correlated with higher the levels of receptive vocabulary. Administered by research assistant to female guardian.
Receptive vocabulary assessment at 12 months | 12 months
  Assess Receptive vocabulary based on the Preschool Language Scale-5 (PLS-5) 5th Edition Parent Questionnaire. The scale accesses: Total language, auditory comprehension, expressive communication standard scores, growth scores, percentile ranks, language age equivalents. PLS-5 scores range anywhere from 40-160 with the mean being 100 and an SD of 15. Higher percentile ranks are correlated with higher the levels of receptive vocabulary. Administered by research assistant to female guardian.
Receptive vocabulary assessment at 24 months | 24 months
  Assess Receptive vocabulary based on the Preschool Language Scale-5 (PLS-5) 5th Edition Parent Questionnaire. The scale accesses: Total language, auditory comprehension, expressive communication standard scores, growth scores, percentile ranks, language age equivalents. PLS-5 scores range anywhere from 40-160 with the mean being 100 and an SD of 15. Higher percentile ranks are correlated with higher the levels of receptive vocabulary. Administered by research assistant to female guardian.

SECONDARY OUTCOMES:
Parental behavior at 12 months | 12 months
  StimQ is an interview-based instrument to assess the family cognitive environment. StimQ-Infant has four scale scores, which add up to the total StimQ Score. ALM Scale ranges 0-6, READING Scale Score ranges 0-15, PIDA Scale Score ranges 0-7, and PVR Scale Score ranges 0-11. The highest total StimQ Score is 39 and the lowest is 0. Higher StimQ scores are correlated with better parental behavior. StimQ-Infant will be done up to 15 months. Administered by research assistant to female guardian.
Parental behavior at 24 months | 24 months
  StimQ is an interview-based instrument to assess the family cognitive environment. StimQ-toddler has four scale scores, which add up to the total StimQ Score. ALM Scale ranges 0-7, READING Scale Score ranges 0-18, PIDA Scale Score ranges 0-10, and PVR Scale Score ranges 0-4. The highest total StimQ Score is 39 and the lowest is 0.Higher StimQ scores are correlated with better parental behavior. StimQ-Toddler will be done up to 27 months. Administered by research assistant to female guardian.

OTHER OUTCOMES:
Child socio-emotional development at 3 months | 3 months
  The Ages and Stages Questionnaire (ASQ) is a questionnaire completed by parents to identify and screen for social and emotional behaviors in their children. The ASQ questionnaire has measures child behaviors and emotional responses assessing seven different areas: self-regulation, compliance, social-communication, adaptive functioning, autonomy, affect, and interaction with people. the questionnaire uses a point system per question that ranges from 0-10. The total score ranges from 0-110+. Total child scores ranging from 0-50 results in "no or low risk" and means the child's social-emotional development appears to be on schedule. Total child scores ranging from 50-65 results in "monitoring" and means child's behavior of concern need to be monitored. Total child scores ranging from 65-110+ results in "refer" and means further assessment with a professional may be needed. Administered by research assistant to female guardian.
Child socio-emotional development at 12 months | 12 months
  The Ages and Stages Questionnaire (ASQ) is a questionnaire completed by parents to identify and screen for social and emotional behaviors in their children. The ASQ questionnaire has measures child behaviors and emotional responses assessing seven different areas: self-regulation, compliance, social-communication, adaptive functioning, autonomy, affect, and interaction with people. the questionnaire uses a point system per question that ranges from 0-10. The total score ranges from 0-110+. Total child scores ranging from 0-50 results in "no or low risk" and means the child's social-emotional development appears to be on schedule. Total child scores ranging from 50-65 results in "monitoring" and means child's behavior of concern need to be monitored. Total child scores ranging from 65-110+ results in "refer" and means further assessment with a professional may be needed. Administered by research assistant to female guardian.
Child socio-emotional development at 24 months | 24 months
  The Ages and Stages Questionnaire (ASQ) is a questionnaire completed by parents to identify and screen for social and emotional behaviors in their children. The ASQ questionnaire has measures child behaviors and emotional responses assessing seven different areas: self-regulation, compliance, social-communication, adaptive functioning, autonomy, affect, and interaction with people. the questionnaire uses a point system per question that ranges from 0-10. The total score ranges from 0-110+. Total child scores ranging from 0-50 results in "no or low risk" and means the child's social-emotional development appears to be on schedule. Total child scores ranging from 50-65 results in "monitoring" and means child's behavior of concern need to be monitored. Total child scores ranging from 65-110+ results in "refer" and means further assessment with a professional may be needed. Administered by research assistant to female guardian.
Parenting Stress at 3 months | 3 months
  The Parenting Stress Index (PSI) is a questionnaire completed by parents designed to measure the magnitude of stress in a parent-child system, to identify dysfunctional parenting with the potential for parental behavioral problems and child adjustment difficulties.The 36-item form includes three subscales: parental distress, parent-child dysfunctional interaction, and difficult child. Coefficient alpha reliability is 0.80-0.87 for the subscales and 0.91 for the total scale. Six-month test-retest reliability is 0.84.
Parenting Stress at 12 months | 12 months
  The Parenting Stress Index (PSI) is a questionnaire completed by parents designed to measure the magnitude of stress in a parent-child system, to identify dysfunctional parenting with the potential for parental behavioral problems and child adjustment difficulties.The 36-item form includes three subscales: parental distress, parent-child dysfunctional interaction, and difficult child. Coefficient alpha reliability is 0.80-0.87 for the subscales and 0.91 for the total scale. Six-month test-retest reliability is 0.84.
Parenting Stress at 24 months | 24 months
  The Parenting Stress Index (PSI) is a questionnaire completed by parents designed to measure the magnitude of stress in a parent-child system, to identify dysfunctional parenting with the potential for parental behavioral problems and child adjustment difficulties.The 36-item form includes three subscales: parental distress, parent-child dysfunctional interaction, and difficult child. Coefficient alpha reliability is 0.80-0.87 for the subscales and 0.91 for the total scale. Six-month test-retest reliability is 0.84.

CONTACTS AND LOCATIONS:
Overall Officials: Renee Boynton, MD, ScD, Principal Investigator — Boston Medical Center
Locations (1):
- Boston Medical Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No